CLINICAL TRIAL: NCT03728738
Title: Zero Degree Head Positioning in Hyperacute Large Artery Ischemic Stroke
Acronym: ZODIAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Anne Alexandrov, Professor of Nursing & Professor of Neurology, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01NR017850-01 (NIH); 1R01NR017850-01 (NIH)
Record Dates: First submitted 2018-10-23; First posted 2018-11-02 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Prospective randomized open blinded endpoint (PROBE) clinical trial using clinical assessors blinded to the intervention to determine neurologic deterioration on the NIH Stroke Scale Score following positioning to either zero degree or thirty degree heights.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero Degree HOB (Experimental): Randomization to zero degree head of bed positioning until the time of initiation of thrombectomy
  Interventions: Procedure: Head of Bed Positioning
- Thirty Degree HOB (Active Comparator): Randomization to thirty degree head of bed positioning until the time of initiation of thrombectomy
  Interventions: Procedure: Head of Bed Positioning

INTERVENTIONS:
Procedure: Head of Bed Positioning — The head of bed (HOB) position will be selected through computerized randomization, and will include either zero degree positioning or thirty degree HOB elevation

SUMMARY:
Placing the head of bed (HOB) at 0-degrees has been shown in small studies to improve blood flow to the brain in patients with ischemic stroke caused by large artery occlusions, thereby reducing stroke symptom worsening. This simple yet potentially impactful intervention has yet to be tested in a large clinical trial in hyperacute large artery ischemic stroke patients, but may provide nurses with a powerful contribution to acute stroke care that is capable of preventing worsening of stroke symptoms and promoting stabilization. Because stroke is the leading cause of preventable long-term disability in adults, this study may show that simple methods such as 0-degree HOB positioning should be considered one of the very first actions taken in the emergent management of acute ischemic stroke patients.

DETAILED DESCRIPTION:
Positioning of the patient during hyperacute ischemic stroke (AIS) treatment is an important, yet understudied aspect of nursing care that could impact the course of treatment and clinical outcome. Since 1968, clinical symptom worsening in AIS patients has been documented with the head of bed (HOB) elevated to 30 degrees or higher, while clinical improvement or symptom stability has been noted with zero degree HOB positioning. Mechanisms for zero degree HOB clinical improvement include favorable gravitational blood flow conditions and recruitment of collateral blood channels, while in the case of treatment with clot-busting medications, increased blood flow may allow more medication to reach occluded arteries facilitating clot breakdown. Despite this, there is currently divide within the clinical community about what position is best for patients, although it has been argued that zero degree head positioning should be among the first steps taken to improve blood flow to the brain and prevent stroke symptom worsening. The investigators have shown that elevated ICP is absent in early AIS, and that pneumonia is rare using these piloted methods. However, no large clinical trial has examined efficacy and safety of zero degree HOB positioning within hyperacute large vessel occlusion (LVO) ischemic stroke patients with potentially viable brain tissue, leaving the acute stroke community confused as to what constitutes best practice. ZODIAC is a prospective randomized open blinded endpoint (PROBE) clinical trial of head positioning to determine if zero degree HOB positioning during the early phase of hyperacute LVO ischemic stroke management prevents neurological symptom worsening. Mechanical thrombectomy (MT) eligible patients (n=182) will be randomized to one of two groups: 1) Zero degree HOB positioning; or, 2) thirty degree HOB positioning. The hypothesis is that optimal HOB position can be determined by early neurological symptom worsening during the intervention (Aim 1) prior to initiation of the thrombectomy procedure, and the investigators propose that real-time deterioration may be a surrogate measure for decreased downstream perfusion, potentially impacting viability of brain at risk for infarction. Aim 2 will confirm that use of zero degree HOB positioning for AIS is safe. Use of this nursing measure holds significant promise as an innovative adjunct method to improve AIS symptoms, and ultimately reduce disability.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke symptoms consistent with large artery occlusion
* Baseline standard of care non-contrast head CT (or MRI) negative for hemorrhage or mass-effect
* Evidence of arterial occlusion on standard of care CT angiography or MR angiography
* Favorable neuroimaging (Alberta Stroke Program Early Computed Tomography Score [ASPECTS] > 6 in anterior circulation stroke; not applicable in posterior circulation stroke)
* Ordered treatment with mechanical thrombectomy
* Pre-stroke baseline modified Rankin Score (mRS) < 1
* Ability to enroll, randomize and begin the intervention within the Emergency Department

Exclusion Criteria:

* Non-English speaking subjects will be excluded due to use of English language instruments (modified Rankin Scale [mRS] & NIHSS) and English speaking investigators
* Pregnancy or suspicion of pregnancy
* Evidence or suspicion of vomiting any time prior to consent which could predispose to aspiration pneumonia and therefore confound determination of protocol safety
* Anticipated palliative care referral
* Evidence of evolving malignant infarction on admission noncontrast CT (or MRI)
* Need for intubation with mechanical ventilation, or non-invasive ventilatory support with either bi-level positive airway pressure (BiPAP) or continuous positive airway pressure (CPAP)
* Inability to tolerate zero-degree positioning due to congestive heart failure, preexisting pneumonia, chronic obstructive pulmonary disease, or other medical condition
* Admission chest radiograph positive for pleural effusion, pulmonary edema, pneumonia, or other pulmonary condition that may confound determination of protocol safety
* Abnormal breath sounds on admission assessment that may confound determination of protocol safety
* Lack of a telephone and/or permanent address predisposing patients to be lost to follow up
* Enrollment in another clinical trial that may affect our primary or secondary endpoints
* In the absence of a consenting legal next of kin, any medical, psychological, cognitive, social or legal condition that would interfere with informed consent and/or capacity to comply with all study requirements, including the necessary time commitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Early Neurologic Deterioration (END) on the National Institute of Health Stroke Scale Occurring During the Positioning Intervention | Measured every 10 minutes from initiation of positioning up until thrombectomy commences or 2 hours - whichever comes first
  Two or more point-worsening in the National Institute of Health Stroke Scale (stroke disability severity measure, ranging from 0-no disability, to 42-severely disabled) score during the positioning intervention period.

SECONDARY OUTCOMES:
Severe Neurological Deterioration (SND) on the National Institute of Health Stroke Scale Occurring During the Positioning Intervention | Measured every 10 minutes from initiation of positioning up until thrombectomy commences or 2 hours - whichever comes first
  Four or more point-worsening in the National Institute of Health Stroke Scale (stroke disability severity measure, ranging from 0-no disability, to 42-severely disabled) score during the positioning intervention period.
Diagnosis of Pneumonia Made During Hospitalization in a Patient Free From Pneumonia at Time of Hospital Admission | Measured up until hospital discharge or day 7 (whichever comes first)
  Documented onset of a new or progressive infiltrate on pulmonary imaging along with the presence of at least two of the following - Fever of 38°C/100.4°F; Purulent sputum; Leukocytosis or leukopenia; and/or, Decline in oxygen saturation.
Participant Deaths within 90-days from Stroke Onset | Up until 90-days from stroke onset
  All cause death occurring from time of randomization up until 90-days from stroke onset
National Institutes of Health Stroke Scale Score at Hospital Discharge or Day 7 | Measured at hospital discharge or by day 7 (whichever comes first)
  Total National Institute of Health Stroke Scale (stroke disability severity measure, ranging from 0-no disability, to 42-severely disabled) score measured at the time of hospital discharge or on day 7
Modified Rankin Scale Score at Hospital Discharge or Day 7 | Measured at hospital discharge or on day 7 (whichever comes first)
  Categorical rank on the Modified Rankin Scale score (stroke functional outcome measure ranging from 0-no functional disability, to 6-dead) measured at the time of hospital discharge or on day 7 (whichever comes first)
Modified Rankin Scale Score at 90-days from Stroke Onset | Measured at 90 days from Stroke Onset
  Categorical rank on the Modified Rankin Scale score (stroke functional outcome measure ranging from 0-no functional disability, to 6-dead) measured at 90 days from stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Anne W Alexandrov, PhD, Principal Investigator — University of Tennessee Health Science Center at Memphis
Locations (11):
- United States (11):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Doctors Medical Center, Modesto, California
  - Northwestern Central DuPage Hospital, Winfield, Illinois
  - University of Louisville Hospital, Louisville, Kentucky
  - Moses Cone Medical Center, Greensboro, North Carolina
  - Saint Francis Health System, Tulsa, Oklahoma
  - Hershey Medical Center - Penn State Health, Hershey, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - Medical City - Fort Worth, Fort Worth, Texas
  - Memorial Hermann Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alexandrov AW, Shearin AJ, Mandava P, Torrealba-Acosta G, Elangovan C, Krishnaiah B, Nearing K, Robinson E, Guthrie-Chu C, Holzmann M, Fill B, Trivedi DR, Richardson A, Middleton S, Brewer BB, Liebeskind DS, Goyal N, Grotta JC, Alexandrov AV; ZODIAC Investigators. Optimal Head-of-Bed Positioning Before Thrombectomy in Large Vessel Occlusion Stroke: A Randomized Clinical Trial. JAMA Neurol. 2025 Sep 1;82(9):905-914. doi: 10.1001/jamaneurol.2025.2253. PMID 40465238